CLINICAL TRIAL: NCT06622785
Title: Examination of the Perceptions of Benefits and Obstacles Related to Physical Activity of Participants in Different Age Groups
Brief Title: Physical Activity of Participants in Different Age Groups
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 06.10.2022-1089
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Adults 18 Years and Older (no Other Exclusion Criteria)
Keywords: healthy; people; physical activity; age
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (3):
- Group 1: People aged 18-29 years
  Interventions: Behavioral: Physical activity; Behavioral: Exercise Benefits
- Group 2: People aged 30-44 years
  Interventions: Behavioral: Physical activity; Behavioral: Exercise Benefits
- Group 3: People aged 45-60 years
  Interventions: Behavioral: Physical activity; Behavioral: Exercise Benefits

INTERVENTIONS:
Behavioral: Physical activity — Data were collected using a International Physical Activity Questionnaire-Short Form (IPAQ-SF)
Behavioral: Exercise Benefits — Data were collected using a Exercise Benefits/Barriers Scale .

SUMMARY:
The subject of the research is to determine the physical activity levels of the participants in different age categories and to determine and analyse participants' perceptions of the benefits of physical activity and the factors that prevent from doing physical activity.

DETAILED DESCRIPTION:
The subject of the research is to determine the physical activity levels of the participants in different age categories and to determine and analyse participants' perceptions of the benefits of physical activity and the factors that prevent from doing physical activity. In this study, it is aimed to determine the physical activity levels of individuals in different age categories and to determine the barriers and benefit perceptions of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old

Exclusion Criteria:

* Not volunteering for research
* Those with incomplete evaluation forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty people
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Descriptive assessment | Baseline
  In the descriptive information form (age, gender, weight, height, etc.) were questioned and recorded.
Exercise benefits and barriers | baseline
  The scale is a 4-point Likert-type and consists of 43 items. It has two subgroups: the benefit scale (29 questions) and the barrier scale (14 questions). A high total score on the scale shows how much the individual believes in exercise.
Physical activity | baseline
  The International Physical Activity Questionnaire-Short Form is a valid and reliable questionnaire to determine physical activity levels in the health and daily lives of adults. It consists of 7 questions evaluating how much PA they have performed in the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Demirtaş, Msc, Principal Investigator — Niğde Ömer Halisdemir University; Arife Akbulut Bayrak, Msc, Principal Investigator — Ankara Yildirim Beyazıt University; Havva Sümeyye Eroğlu, Msc, Principal Investigator — Gazi University
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared with third parties. The informed consent form has been prepared and approved in this way.